CLINICAL TRIAL: NCT06344182
Title: Reliability, Concurrent Validity and Minimal Detectable Change of the Step Up and Down Test in Patients With Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sumeyya Tarkan, Pt, Dokuz Eylul University
Other Study IDs: STarkan
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; stair climbing; reliability; validity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Step Up and Down Test — Step Up and Down Test In the StUD test, the patient completes maximum number of step-up-down repetitions in 15 seconds. Starting from a standing position, the participant took a full step up, leading with the test leg, then the non-testing leg, until both knees were fully extended and both hips were at least in neutral extension. In order to stress the testing limb concentrically and eccentrically, the participant stepped off the step first with the non-testing limb, then the testing limb. The patient was asked to repeat for 15 seconds as quickly as possible. The physical therapist stood to the side of the step for safety and so that he/she could observe the technique and ensure that the participant came to a full step up and down during the test.

SUMMARY:
The aim of the study is to measure the validity and reliability of the StUD test in patients with TKA. Forty-seven patients with primary TKA included in this study. The test-retest reliability of the StUD test was measured with 1-hour interval. Validity was assessed that the 30s Chair Stand Test (30sCS), the Hospital for Special Surgery score (HSS) and Short Form-12 Quality Life Questionnaire (SF-12) were used as comparator instruments.

DETAILED DESCRIPTION:
The study was designed as test-retest research. This study was approved by the ethics committee of Dokuz Eylul University, Izmir, Turkey. This study was conducted between 2021 and 2022 at the Dokuz Eylul University Hospital Orthopedics Department, Izmir, Turkey. Informed consent was obtained from all participants in accordance with the Declaration of Helsinki.

Sample Size The NCSS Trial and PASS 14 software (NCSS, LLC, Kaysville, Utah USA) was used to conduct the sample size. Power of 0.8 and an alpha level of 0.05 were used. Previous research on StUD in patients with knee Osteoarthritis was noted good test-retest reliability (ICC= 0.87) (G. P. L. Almeida et al., 2021). The test-retest reliability of the current study was thus hypothesized to be excellent. Assuming a %10 attrition rate, a null reliability with ICC=0.75 and expected reliability with ICC=0.90, 47 subjects would be needed.

Participant Forty-seven patients with primary TKA who were operated on by the same surgeon using the paramedian approach were contacted by phone and volunteered to participate in this study. Patients with primary TKA who are at least six months post-surgery were included. Patients were selected and invited to the study by the surgeon and physiotherapist.

Statistical Analysis All data were analyzed using the IBM SPSS Statistics (Version 23.0) software. The Kolmogorov-Smirnov/Shapiro-Wilk tests were used for the determination of the normal distribution. The difference between the pain levels before and after the trials was compared using the Paired Samples T test. The level of significance was determined p < .05. The correlations between the StUD and 30 CST, HSS, PCS12, and MCS12 were calculated to determine convergent validity. The convergent validity was analyzed based on the Spearman's correlation and was interpreted as follows: 0-0.09 = no correlation; 0.1-0.39 = weak correlation; 0.4-0.59 = moderate correlation; 0.7-0.89 = strong correlation; and 0.9-1 = perfect correlation. Paired samples' t test was used for comparing the difference between the first and second trials of StUD test. The intraclass correlation coefficient (ICC2,1) was used assess the test-retest reliability. The ICC values were interpreted as follows: poor, <0.5; moderate, 0.5-0.75; good, 0.75-0.9; excellent reliability, >0.9 (Koo & Li, 2016). The standard error of measurement (SEM) was calculated as SD×√(1-ICC) , where SD is the pooled standard deviation from the first session. Minimal detectable change (MDC) was calculated at a 95% confidence level (MDC95). MDC95 was calculated according to following formula: MDC95=SEM×1.95×√2. All data were analyzed using the IBM SPSS Statistics (Version 23.0) software

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary TKA who are at least six months post-surgery
* Patients over 40 years of age

Exclusion Criteria:

* having a body mass index (BMI) greater than 40 kg/m2,
* having had other surgery on a leg with TKA,
* having symptomatic hip OA,
* having a history of knee or hip fracture,
* having a previous orthopedic or neurological disease that prevents stepping

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary TKA who were operated on by the same surgeon using the paramedian approach were contacted by phone and volunteered to participate in this study. Patients with primary TKA who are at least six months post-surgery were included. Patients were selected and invited to the study by the surgeon and physiotherapist
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Step Up and Down Test | 2021
  In the StUD test, the patient completes maximum number of step-up-down repetitions in 15 seconds.

SECONDARY OUTCOMES:
30 Seconds Chair Stand Test | 2021
  The 30 CST is a valid and reliable performance-based test to assess lower extremity muscle strength in patients with TKA.

OTHER OUTCOMES:
Hospital for Special Surgery (HSS) Knee Score | 2021
  The HSS knee score criteria are based on a total of 100 points. The score consists of seven categories: Pain, function, range of motion, muscle strength, flexion deformity, instability, and subtractions.
12-Item Short-Form Health Survey | 2021
  Health-related quality of life (HRQOL) was assessed with the Short Form Health Survey-12 (SF-12).

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Almeida GJ, Schroeder CA, Gil AB, Fitzgerald GK, Piva SR. Interrater reliability and validity of the stair ascend/descend test in subjects with total knee arthroplasty. Arch Phys Med Rehabil. 2010 Jun;91(6):932-8. doi: 10.1016/j.apmr.2010.02.003. PMID 20510986
- [Background] Almeida GPL, Monteiro IO, Dantas RGO, Tavares MLA, Lima POP. Reliability, validity and responsiveness of the Step Up and Down (StUD) test for individuals with symptomatic knee osteoarthritis. Musculoskelet Sci Pract. 2021 Dec;56:102454. doi: 10.1016/j.msksp.2021.102454. Epub 2021 Sep 1. PMID 34482195
- [Background] Eymir M, Yuksel E, Unver B, Karatosun V. Reliability, validity, and minimal detectable change of the Step Test in patients with total knee arthroplasty. Ir J Med Sci. 2022 Dec;191(6):2651-2656. doi: 10.1007/s11845-021-02888-6. Epub 2022 Jan 13. PMID 35022951
- [Background] Narin S, Unver B, Bakirhan S, Bozan O, Karatosun V. Cross-cultural adaptation, reliability and validity of the Turkish version of the Hospital for Special Surgery (HSS) Knee Score. Acta Orthop Traumatol Turc. 2014;48(3):241-8. doi: 10.3944/AOTT.2014.3109. PMID 24901911